CLINICAL TRIAL: NCT03440216
Title: Population Pharmacokinetics and Pharmacodynamics of Beta-lactams of Interest in Adult Patients From Intensive Care Units
Acronym: Pop-PK/PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Paul M. Tulkens, Professor, Université Catholique de Louvain
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pop PK/PD betalactams ICU
Record Dates: First submitted 2018-01-18; First posted 2018-02-22 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Pharmacokinetics; Anti-Bacterial Agents; Infection, Bacterial; Infections, Respiratory; Infection; Drug Monitoring
Keywords: temocillin; ceftriaxone; meropenem; pharmacokinetics; pharmacodynamics; Intensive Care; dosing; total concentration; free concentration
MeSH Terms: conditions — Bacterial Infections; Respiratory Tract Infections; Infections | interventions — Blood Specimen Collection; temocillin; Ceftriaxone; Meropenem

STUDY DESIGN:
Intervention Model Description: 2 groups of patients studied in parallel
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sampling if GFR = or > 30 mL/min (Experimental): Note: GFR = Glomerular Filtration Rate
  Patients with a normal of moderately decreased renal function
  * Temocillin: 6 g in continuous infusion over 24 h;
  * Ceftriaxone: bolus 2 g (in 30 min) every 12h
  * Meropenem: prolonged infusion (3 h) of 2 g every 8h
  Blood sampling for antibiotic (temocillin, ceftriaxone or meropenem) pharmacokinetic analysis / Tissue sampling (lung) for determination of antibiotic content when possible / Collection of fluid samples (bronchoalveolar lavage, drainage fluid) for determination of antibiotic concentration when possible
  Interventions: Drug: blood sampling; Drug: Tissue sampling (lung); Drug: Collection of fluid samples
- Sampling if GFR < 30 mL/min (Experimental): Patients with severe renal insufficiency or hemodialysis:
  * Temocillin: 6 g in continuous infusion over 24 h;
  * Ceftriaxone: bolus 2 g (in 30 min) every 12h
  * Meropenem: prolonged infusion (3 h) of 2 g every 8h
  Blood sampling for antibiotic (temocillin, ceftriaxone or meropenem) pharmacokinetic analysis / Tissue sampling (lung) for determination of antibiotic content if possible / Collection of fluid samples (bronchoalveolar lavage, drainage fluid) for determination of antibiotic concentration if possible
  Interventions: Drug: blood sampling; Drug: Tissue sampling (lung); Drug: Collection of fluid samples

INTERVENTIONS:
Drug: blood sampling — * temocillin: blood sampling every day for 7 days
  * ceftriaxone: blood sampling 12h after administration for 7 days
  * meropenem: blood sampling at 1h, 3h, 5h and 8h after initiation of the administration at days 1 and 2; one sampling at 8h on days 3 to 7
  Other Names: temocillin, ceftriaxone, meropenem
Drug: Tissue sampling (lung) — Sampling of tissue (lung) when possible during treatment for measurement of the content in antibiotic (temocillin, ceftriaxone, or meropenem, depending on the drug received by the patient)
  Other Names: temocillin, ceftriaxone, meropenem
Drug: Collection of fluid samples — Collection of fluid samples (bronchoalveolar lavage, drainage fluid) for determination of antibiotic ((temocillin, ceftriaxone, or meropenem, depending on the drug received by the patient) concentration when possible during treatment
  Other Names: temocillin, ceftriaxone, meropenem

SUMMARY:
Antibiotics are still most often administered on an empiric fashion, as defined for the general population with dosages only adapted based on weight and renal and/or hepatic functions. As a result, serum concentrations show important interpatient variations with the risk of being subtherapeutic or toxic. Recent studies with temocillin, ceftriaxone, or meropenem confirm this for patients in intensive care units.

The aim of the study will be to measure the total and free concentrations of temocillin, ceftriaxone, and meropenem in patients hospitalized in Intensive Care Units for pulmonary infections or another infection for which one of the above mentioned antibiotics is indicated. Patients will be stratified according to the level of their renal function. The antibiotics will be assayed in plasma as well as other accessible fluids in order to assess their pharmacokinetic properties.

DETAILED DESCRIPTION:
1. Background, Literature Survey and Justification of The Study

   1.1. Introduction

   β-lactams efficacy depends primarily from the time interval during which the plasma concentration remains above the minimal inhibitory concentration (MIC) of the antibiotic against the target organism(s) (Craig, 1998). It is generally accepted that the free concentration of the antibiotic must remain above the MIC for at least 40 to 70% of the interval between two successive administrations, and should even reach 100% for severe infections in patients hospitalized in Intensive Care Units (MacGowan, 2011). The free concentration must reach a value of 4 x the MIC for 40 to 70% (Mohd Hafiz et al., 2012) or even 100 % (Tam et al., 2005) of the dosing interval in order to prevent the emergence of resistance.

   Due to the large inter- and intraindividual variations between patients, it is difficult to reach the desired concentrations if relying only on usual dosage recommendations and/or using standard dosing regimens. Moreover, Intensive Care patients are difficult patients in this context (Roberts et al., 2014) due to gross perturbations related to underlying diseases and abnormalities (arterial hypertension, cardiac rhythm alterations, renal and/or hepatic insufficiency) and the necessary interventions (artificial ventilation, surgery, artificial feeding, and so on…). They also show important variations in the level of plasma proteins and rapid and unpredictable fluctuations of their renal function (Beumier et al., 2015; Goncalves-Pereira and Povoa, 2011; Roberts and Lipman, 2009), all of which are known to modulate the pharmacokinetics of β-lactams (Goncalves-Pereira and Povoa, 2011; Hayashi et al., 2013; Sime et al., 2012; Udy et al., 2012; Wong et al., 2013). The concentration of the free fraction will be especially modified for those β-lactams with large protein binding such as temocillin or ceftriaxone (Schleibinger et al., 2015; Ulldemolins et al., 2011; Van Dalen et al., 1987; Wong et al., 2013), but may also be altered for β-lactams that are mainly excreted via the renal route (temocillin, ceftriaxone, meropenem) (Carlier et al., 2013; Simon et al., 2006; Vandecasteele et al., 2015).

   1.2. Clinical Interest of temocillin, ceftriaxone and meropenem and State of the Art Concerning their dosing

   Temocillin is a carboxypenicillin with useful activity against Gram-negative bacteria (excluding P. aeruginosa) and with a large stability towards most β-lactamases, including ESBL), AmpC cephalosporinases, and some carbapenemases (Livermore et al., 2006; Zykov et al., 2016). Temocillin may stand as an alternative to carbapenems (Balakrishnan et al., 2011; Livermore and Tulkens, 2009). About 85% of temocillin in plasma is protein-bound and about 80% of the administered dose is eliminated in 24 h under an intact form by glomerular filtration and tubular secretion (Temocillin Summary of Product Characteristics [SmPC], 2015)

   Ceftriaxone shows a moderately enlarged spectrum of activity and is stable towards certain β-lactamases but not to ESBLs, AmpC cephalosporinases and certain carbapenemases (Suankratay et al., 2008). It is an alternative to carbapenems when dealing with an infection with susceptible organisms (Paradis et al., 1992). Its protein binding is about 95%, and its elimination is mainly via the renal route (50 to 60% under an unchanged form) with the remaining eliminated via the bile to form microbiologically inactive metabolites (Ceftriaxone SmPC, 2015).

   Meropenem shows a very large spectrum and is used in empiric therapy when fearing the presence of ESBL-producing organisms to which other antibiotics are resistant (Zykov et al., 2016). Meropenem has an unpredictable pharmacokinetic profile in patients with renal insufficiency or under hemodialysis (Carlier et al., 2013; Goncalves-Pereira et al., 2014). Meropenem is mainly excreted via the renal route (50 - 75 % under an unchanged form; SmPC meropenem, 2014).

   Antibiotic are often prescribed empirically with doses based on what has been found appropriate for the general population, with some adaptation for weight and renal and/or hepatic function. As for any drug, however, there is increasing evidence that the concentrations observed after administration of a standard dose are actually highly variable and often different from the expected ones, leading to risks of sub-therapeutic or toxic effects.

   Recent studies have shown that an intravenous administration of 6 g of temocillin by continuous infusion (Laterre et al., 2015), of 4 g of ceftriaxone in two administrations at 12 h interval (Roberts et al., 2007; Salvador et al., 1983), or of 6 g of meropenem in 3 administrations by prolonged infusion (3 h) at 8 h interval (Dulhunty et al., 2013; Frippiat et al., 2015; Jamal et al., 2015), allow to reach free plasma concentrations of 4 x the MIC against susceptible organisms during 40-70%, or even 100% of the dosing interval, with, however, large inter-individual variations, especially for molecules with high protein biding (temocillin, ceftriaxone) due to variations in their renal elimination. Very little information is available about their tissue levels but it is suspected that large inter-individual variations are also frequent.
2. Study Objectives

   The goal is to measure the total and free concentrations of the antibiotics in plasma, accessible body fluids and, if possible, tissues after intravenous administration of:
   * temocillin: 6 g by continuous infusion over 24 h;
   * ceftriaxone: bolus administration of 2 g in a 30 min infusion twice daily;
   * meropenem: prolonged infusion (3 h) of 2 g three times daily.

   These doses will be adjusted in patients based on their renal function.

   Primary objective:

   To calculate and assess the values of key pharmacokinetic parameters (total clearance, volume of distribution, constants of elimination, plasma and tissue total exposure, and maximal and minimal plasma and body fluid concentrations.

   Secondary objectives:
   * the correlation between the plasma protein profile and the actual free antibiotic concentrations;
   * the impact of the alterations of the renal function on the free and total plasma concentrations of the antibiotics;
   * the impact of the level and nature of circulating proteins on the free fraction of the antibiotics;
   * the extent of the tissular penetration of the antibiotics (in accessible samples) and of their penetration in pertinent body fluids (bronchoalveolar lavage, drainage and ascites fluids.
   * to model the population pharmacokinetics of the antibiotics in the whole set of patients included in the study;
   * to investigate and assess the influence of co-variates (using biometric, biochemical and clinical data) on the variability of the individual pharmacokinetic profiles.
3. Outcome measures

   • Primary Outcome Measure: Impact of renal function on total plasma concentrations (Measurement of total plasma antibiotic concentrations)

   • Secondary Outcome Measures:
   * Impact of the plasma protein concentration and of their nature on the free concentration of antibiotics
   * Tissular and fluid penetration of antibiotics (lung tissue, bronchoalveolar lavage, drainage fluids)
   * Pharmacokinetic modeling
   * Co-variates analysis
4. Conduct of the Study

   4.1. Eligible patients

   Patients hospitalized in Intensive Care Units and treated for pulmonary or abdominal infection, septicemia, or any other infection calling for the prescription of one of the three antibiotics mentioned above.

   4.2. Study groups

   Patients will be divided in two groups: :
   * Group 1: patients with a glomerular filtration rate (GFR) ≥ 30 mL/min
   * Group 2: patients with renal insufficiency or under hemodialysis

   4.3. Safety considerations

   The three β-lactams have each a long record of safe use in patients hospitalized in Intensive Care Units but may cause an alteration of the commensal flora, allergic reactions, neurotoxicity (at high doses). Ceftriaxone may case hemolytic anemia.

   4.4. Exclusion criteria
   * Patients of <18 years
   * Allergy to β-lactams
   * Hypersensitivity to penicillin (IgE-mediated)
   * Any biological abnormality considered by the attending physician as susceptible to interfere in a significant manner on the interpretation of the data
   * Absence of consensus
   * Therapeutic limitation

   4.5. Treatment duration: 7 days except for deep, non-controlled foci (extended to 10-14 days).

   4.6. Follow up: First visit (visit #1) to determine eligibility criteria. Additional visits: each day during the treatment period.
5. Calculation of the number of patients

   As this is a descriptive pharmacokinetic study without formal predefined hypothesis, no calculation of the size of the population has been made. Based on literature data and the experience of the investigators, a total of 20 patients in each arm should be sufficient to draw meaningful conclusions.
6. Sampling and processing of samples

   * Sampling of serum and body fluids: typically at equilibrium for all three antibiotics, and at fixed times after administration of the bolus (ceftriaxone) or the prolonged infusion (meropenem), and performed by a research nurse according to a predefined schedule.
   * Sampling of tissues: by Medical personnel when justified for diagnostic or treatment reasons.
   * All samples will transferred to the laboratory where they will be treated using predefined and validated protocols.

   Antibiotic assay: validated liquid chromatography - mass spectrometry methods (protocols and performance of the assay methods available upon request). The free fraction of each antibiotic will be measured after separation of the bound fraction by molecular sieving (Ngougni Pokem et al., 2015).
7. Statistical analysis and data analysis

   Pharmacokinetic analyses will be performed using either NONMEM (NONlinear Mixed Effect Modeling) (http://www.iconplc.com/innovation/nonmem/ ) or PMETRICS (http://www.lapk.org/pmetrics.php) software. Mono-, bi-, and tri-compartmental models will be tested using plasma, tissular and body fluids antibiotic free and total antibiotic concentrations. The First-Order Conditional Estimation with Interaction (FOCE-I) method will be used to assess the objective functions (Jaruratanasirikul et al., 2015) in order to select the most appropriate model for the calculation of the pharmacokinetic parameters (Roberts et al. 2009).
8. Confidentiality and Rights of patients.

   The identity and the personal data of the patients will remain confidential according to the applicable Belgian Law

   Before enrollment, each patient (or his/her guardian) will provide a written informed consent. Each enrolled patients (or his/her guardian) will be allowed to withdraw from the study at any time without impact on his/her treatment.
9. Contacts

All questions concerning the study can be addressed to

* the responsible investigator: Professor Pr Pierre-François Laterre (phone: 00-32-2-764- 2733 (Intensive Care Unit) or 764-2735 (direct) at the Cliniques universitaire St Luc, Brussels, Belgium
* the associated investigators: Professor Françoise Van Bambeke (phone: 00-32-2-764-7378) and Pharm. Perrin Ngougni Pokem (phone 00-32-2-764-7225) at the Université catholique de Louvain (Louvain Drug Research Institute), Brussels, Belgium.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspicion or documentation of of an infection requiring intravenous antibiotic therapy (this includes any patient admitted to the Intensive Care Unit for an infection (or developing an infection) that calls for administration of temocillin, ceftriaxone or meropenem).

Exclusion Criteria:

* Patients allergic to β-lactams
* IgE-mediated hypersensibility to penicillins
* any biological abnormality that the attending physician considers as susceptible to delay or perturb in a significant manner the interpretation of the trial
* lack of accepted informed consent
* patient with therapeutic limitations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Impact of renal function on total plasma concentrations | 36 months
  Measurement of total plasma antibiotic concentrations (measurement by a validated HPLC-MS-MS after suitable extraction; no predefined value set [exploratory])

SECONDARY OUTCOMES:
Impact of the plasma protein concentration and of their nature on the free concentration of antibiotics | 36 months
  Measurement of antibiotic plasma free concentrations and analysis of plasma protein profiles (measurement by a validated HPLC-MS-MS after suitable extraction; no predefined value set [exploratory])
Tissular and fluid penetration of antibiotics (total) | 36 months
  Measurement of total concentrations of antibiotics in tissue samples and fluids (bronchoalveolar lavage, drainage fluids) when obtained (measurement by a validated HPLC-MS-MS after suitable extraction; no predefined value set [exploratory])
Tissular and fluid penetration of antibiotics (free) | 36 months
  Measurement of free concentrations of antibiotics in tissue samples and fluids (bronchoalveolar lavage, drainage fluids) when obtained (measurement by a validated HPLC-MS-MS after suitable extraction; no predefined value set [exploratory])
Pharmacokinetic analysis and population pharmacokinetics: Cmax (total and free) | 36 months
  Analysis of the antibiotic pharmacokinetic profiles by means of appropriate software to calculate the actual mean and median values of the total and free plasma Cmax of temocillin (in mg/L) in the study population and to determine their value in a simulated population (Monte Carlo simulations; 1000 simulated patients)
Pharmacokinetic analysis and population pharmacokinetics: Cmin (total and free) | 36 months
  Analysis of the antibiotic pharmacokinetic profiles by means of appropriate software to calculate the actual mean and median values of the total and free plasma Cmin of temocillin (in mg/L) in the study population and to determine their values in a simulated population (Monte Carlo simulations; 1000 simulated patients)
Pharmacokinetic analysis and population pharmacokinetics: time above a critical concentration value for total and free concentrations | 36 months
  Analysis of the antibiotic pharmacokinetic profiles by means of appropriate software to calculate the actual mean and median values of the fraction of the time between two successive drug administrations during which the total and free plasma concentrations of temocillin remain above a critical value ( "S" breakpoint of the corresponding antibiotic [temocillin: British Society of Antimicrobial Chemotherapy [BSAC] or Belgian Summary of Product Characteristics [SmPC] value; ceftriaxone and meropenem: European Committee for Antimicrobials Susceptibility Testing [EUCAST] value]) in the study population, and to determine its value in a simulated population (Monte Carlo simulations; 1000 simulated patients)
Covariables analysis: biometric values: weight | 36 months
  Assessment of the impact of patient's weight [in kg]
Covariables analysis: biometric values: height | 36 months
  Assessment of the impact of patient's height [in cm]
Covariables analysis: biometric values: age | 36 months
  Assessment of the impact of patient's age [in years]
Covariables analysis: biochemical data: serum total protein and albumin | 36 months
  Assessment of the impact of total serum protein [in g/L] and total serum albumin [in g/L].
Covariables analysis: biochemical data: elevation hepatic transaminases | 36 months
  Assessment of the impact the elevation of the hepatic transaminases [in international units/L, with reference fo the local normal values]
Covariables analysis: biochemical data: blood urea and creatinine | 36 months
  Assessment of the impact of the urea [in mol/L] and creatinine [in mg/L]) blood levels
Covariable analysis: clinical status with respect to infection | 36 months
  clinical status of the patient (in 3 categories: moderately severe infection; severe infection; life-threatening infection) as per the judgment of the attending physician
Covariable analysis: renal function | 36 months
  renal function based on calculated glomerular filtration with a dichotomic cut-off at < 30 ml/min or above

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-François Laterre, MD, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available.

REFERENCES:
- [Result] Goncalves-Pereira J, Silva NE, Mateus A, Pinho C, Povoa P. Assessment of pharmacokinetic changes of meropenem during therapy in septic critically ill patients. BMC Pharmacol Toxicol. 2014 Apr 14;15:21. doi: 10.1186/2050-6511-15-21. PMID 24731745
- [Result] Hayashi Y, Lipman J, Udy AA, Ng M, McWhinney B, Ungerer J, Lust K, Roberts JA. beta-Lactam therapeutic drug monitoring in the critically ill: optimising drug exposure in patients with fluctuating renal function and hypoalbuminaemia. Int J Antimicrob Agents. 2013 Feb;41(2):162-6. doi: 10.1016/j.ijantimicag.2012.10.002. Epub 2012 Nov 13. PMID 23153962
- [Result] Huttner A, Harbarth S, Hope WW, Lipman J, Roberts JA. Therapeutic drug monitoring of the beta-lactam antibiotics: what is the evidence and which patients should we be using it for? J Antimicrob Chemother. 2015 Dec;70(12):3178-83. doi: 10.1093/jac/dkv201. Epub 2015 Jul 17. PMID 26188037
- [Result] Jamal JA, Mat-Nor MB, Mohamad-Nor FS, Udy AA, Wallis SC, Lipman J, Roberts JA. Pharmacokinetics of meropenem in critically ill patients receiving continuous venovenous haemofiltration: a randomised controlled trial of continuous infusion versus intermittent bolus administration. Int J Antimicrob Agents. 2015 Jan;45(1):41-5. doi: 10.1016/j.ijantimicag.2014.09.009. Epub 2014 Oct 18. PMID 25455853
- [Result] Jaruratanasirikul S, Thengyai S, Wongpoowarak W, Wattanavijitkul T, Tangkitwanitjaroen K, Sukarnjanaset W, Jullangkoon M, Samaeng M. Population pharmacokinetics and Monte Carlo dosing simulations of meropenem during the early phase of severe sepsis and septic shock in critically ill patients in intensive care units. Antimicrob Agents Chemother. 2015;59(6):2995-3001. doi: 10.1128/AAC.04166-14. Epub 2015 Mar 9. PMID 25753628
- [Result] Kiem S, Schentag JJ. Interpretation of antibiotic concentration ratios measured in epithelial lining fluid. Antimicrob Agents Chemother. 2008 Jan;52(1):24-36. doi: 10.1128/AAC.00133-06. Epub 2007 Sep 10. No abstract available. PMID 17846133
- [Result] Laterre PF, Wittebole X, Van de Velde S, Muller AE, Mouton JW, Carryn S, Tulkens PM, Dugernier T. Temocillin (6 g daily) in critically ill patients: continuous infusion versus three times daily administration. J Antimicrob Chemother. 2015 Mar;70(3):891-8. doi: 10.1093/jac/dku465. Epub 2014 Nov 27. PMID 25433006
- [Result] Livermore DM, Hope R, Fagan EJ, Warner M, Woodford N, Potz N. Activity of temocillin against prevalent ESBL- and AmpC-producing Enterobacteriaceae from south-east England. J Antimicrob Chemother. 2006 May;57(5):1012-4. doi: 10.1093/jac/dkl043. Epub 2006 Mar 10. No abstract available. PMID 16531428
- [Result] Livermore DM, Tulkens PM. Temocillin revived. J Antimicrob Chemother. 2009 Feb;63(2):243-5. doi: 10.1093/jac/dkn511. Epub 2008 Dec 18. PMID 19095679
- [Result] MacGowan A. Revisiting Beta-lactams - PK/PD improves dosing of old antibiotics. Curr Opin Pharmacol. 2011 Oct;11(5):470-6. doi: 10.1016/j.coph.2011.07.006. Epub 2011 Aug 19. PMID 21862409
- [Result] Martin C, Ragni J, Lokiec F, Guillen JC, Auge A, Pecking M, Gouin F. Pharmacokinetics and tissue penetration of a single dose of ceftriaxone (1,000 milligrams intravenously) for antibiotic prophylaxis in thoracic surgery. Antimicrob Agents Chemother. 1992 Dec;36(12):2804-7. doi: 10.1128/AAC.36.12.2804. PMID 1482149
- [Result] McWhinney BC, Wallis SC, Hillister T, Roberts JA, Lipman J, Ungerer JP. Analysis of 12 beta-lactam antibiotics in human plasma by HPLC with ultraviolet detection. J Chromatogr B Analyt Technol Biomed Life Sci. 2010 Jul 15;878(22):2039-43. doi: 10.1016/j.jchromb.2010.05.027. Epub 2010 May 24. PMID 20561826
- [Result] Mohd Hafiz AA, Staatz CE, Kirkpatrick CM, Lipman J, Roberts JA. Continuous infusion vs. bolus dosing: implications for beta-lactam antibiotics. Minerva Anestesiol. 2012 Jan;78(1):94-104. Epub 2011 Jul 6. PMID 21730935
- [Result] Ngougni Pokem P, Miranda Bastos AC, Tulkens PM, Wallemacq P, Van Bambeke F, Capron A. Validation of a HPLC-MS/MS assay for the determination of total and unbound concentration of temocillin in human serum. Clin Biochem. 2015 May;48(7-8):542-5. doi: 10.1016/j.clinbiochem.2015.02.006. Epub 2015 Feb 21. PMID 25712752
- [Result] Paradis D, Vallee F, Allard S, Bisson C, Daviau N, Drapeau C, Auger F, LeBel M. Comparative study of pharmacokinetics and serum bactericidal activities of cefpirome, ceftazidime, ceftriaxone, imipenem, and ciprofloxacin. Antimicrob Agents Chemother. 1992 Oct;36(10):2085-92. doi: 10.1128/AAC.36.10.2085. PMID 1444289
- [Result] Roberts JA, Abdul-Aziz MH, Lipman J, Mouton JW, Vinks AA, Felton TW, Hope WW, Farkas A, Neely MN, Schentag JJ, Drusano G, Frey OR, Theuretzbacher U, Kuti JL; International Society of Anti-Infective Pharmacology and the Pharmacokinetics and Pharmacodynamics Study Group of the European Society of Clinical Microbiology and Infectious Diseases. Individualised antibiotic dosing for patients who are critically ill: challenges and potential solutions. Lancet Infect Dis. 2014 Jun;14(6):498-509. doi: 10.1016/S1473-3099(14)70036-2. Epub 2014 Apr 24. PMID 24768475
- [Result] Roberts JA, Lipman J. Pharmacokinetic issues for antibiotics in the critically ill patient. Crit Care Med. 2009 Mar;37(3):840-51; quiz 859. doi: 10.1097/CCM.0b013e3181961bff. PMID 19237886
- [Result] Roberts JA, Boots R, Rickard CM, Thomas P, Quinn J, Roberts DM, Richards B, Lipman J. Is continuous infusion ceftriaxone better than once-a-day dosing in intensive care? A randomized controlled pilot study. J Antimicrob Chemother. 2007 Feb;59(2):285-91. doi: 10.1093/jac/dkl478. Epub 2006 Nov 28. PMID 17135183
- [Result] Roberts JA, Kirkpatrick CM, Roberts MS, Robertson TA, Dalley AJ, Lipman J. Meropenem dosing in critically ill patients with sepsis and without renal dysfunction: intermittent bolus versus continuous administration? Monte Carlo dosing simulations and subcutaneous tissue distribution. J Antimicrob Chemother. 2009 Jul;64(1):142-50. doi: 10.1093/jac/dkp139. Epub 2009 Apr 27. PMID 19398460
- [Result] Salvador P, Smith RG, Weinfeld RE, Ellis DH, Bodey GP. Clinical pharmacology of ceftriaxone in patients with neoplastic disease. Antimicrob Agents Chemother. 1983 Apr;23(4):583-8. doi: 10.1128/AAC.23.4.583. PMID 6305263
- [Result] Schleibinger M, Steinbach CL, Topper C, Kratzer A, Liebchen U, Kees F, Salzberger B, Kees MG. Protein binding characteristics and pharmacokinetics of ceftriaxone in intensive care unit patients. Br J Clin Pharmacol. 2015 Sep;80(3):525-33. doi: 10.1111/bcp.12636. Epub 2015 Jun 11. PMID 25808018
- [Result] Sime FB, Roberts MS, Peake SL, Lipman J, Roberts JA. Does Beta-lactam Pharmacokinetic Variability in Critically Ill Patients Justify Therapeutic Drug Monitoring? A Systematic Review. Ann Intensive Care. 2012 Jul 28;2(1):35. doi: 10.1186/2110-5820-2-35. PMID 22839761
- [Result] Simon N, Dussol B, Sampol E, Purgus R, Brunet P, Lacarelle B, Berland Y, Bruguerolle B, Urien S. Population pharmacokinetics of ceftriaxone and pharmacodynamic considerations in haemodialysed patients. Clin Pharmacokinet. 2006;45(5):493-501. doi: 10.2165/00003088-200645050-00004. PMID 16640454
- [Result] Suankratay C, Jutivorakool K, Jirajariyavej S. A prospective study of ceftriaxone treatment in acute pyelonephritis caused by extended-spectrum beta-lactamase-producing bacteria. J Med Assoc Thai. 2008 Aug;91(8):1172-81. PMID 18788687
- [Result] Tam VH, Schilling AN, Neshat S, Poole K, Melnick DA, Coyle EA. Optimization of meropenem minimum concentration/MIC ratio to suppress in vitro resistance of Pseudomonas aeruginosa. Antimicrob Agents Chemother. 2005 Dec;49(12):4920-7. doi: 10.1128/AAC.49.12.4920-4927.2005. PMID 16304153
- [Result] Udy AA, Varghese JM, Altukroni M, Briscoe S, McWhinney BC, Ungerer JP, Lipman J, Roberts JA. Subtherapeutic initial beta-lactam concentrations in select critically ill patients: association between augmented renal clearance and low trough drug concentrations. Chest. 2012 Jul;142(1):30-39. doi: 10.1378/chest.11-1671. PMID 22194591
- [Result] Ulldemolins M, Roberts JA, Rello J, Paterson DL, Lipman J. The effects of hypoalbuminaemia on optimizing antibacterial dosing in critically ill patients. Clin Pharmacokinet. 2011 Feb;50(2):99-110. doi: 10.2165/11539220-000000000-00000. PMID 21142293
- [Result] Van Dalen R, Vree TB, Baars IM. Influence of protein binding and severity of illness on renal elimination of four cephalosporin drugs in intensive-care patients. Pharm Weekbl Sci. 1987 Apr 24;9(2):98-103. doi: 10.1007/BF01960743. PMID 3588249
- [Result] Vandecasteele SJ, Miranda Bastos AC, Capron A, Spinewine A, Tulkens PM, Van Bambeke F. Thrice-weekly temocillin administered after each dialysis session is appropriate for the treatment of serious Gram-negative infections in haemodialysis patients. Int J Antimicrob Agents. 2015 Dec;46(6):660-5. doi: 10.1016/j.ijantimicag.2015.09.005. Epub 2015 Oct 9. PMID 26603304
- [Result] Verdier MC, Tribut O, Tattevin P, Le Tulzo Y, Michelet C, Bentue-Ferrer D. Simultaneous determination of 12 beta-lactam antibiotics in human plasma by high-performance liquid chromatography with UV detection: application to therapeutic drug monitoring. Antimicrob Agents Chemother. 2011 Oct;55(10):4873-9. doi: 10.1128/AAC.00533-11. Epub 2011 Jul 25. PMID 21788467
- [Result] Wong G, Briscoe S, Adnan S, McWhinney B, Ungerer J, Lipman J, Roberts JA. Protein binding of beta-lactam antibiotics in critically ill patients: can we successfully predict unbound concentrations? Antimicrob Agents Chemother. 2013 Dec;57(12):6165-70. doi: 10.1128/AAC.00951-13. Epub 2013 Sep 30. PMID 24080664
- [Result] Zykov IN, Sundsfjord A, Smabrekke L, Samuelsen O. The antimicrobial activity of mecillinam, nitrofurantoin, temocillin and fosfomycin and comparative analysis of resistance patterns in a nationwide collection of ESBL-producing Escherichia coli in Norway 2010-2011. Infect Dis (Lond). 2016 Feb;48(2):99-107. doi: 10.3109/23744235.2015.1087648. Epub 2015 Sep 28. PMID 26414659
- See also: Ceftriaxone. Ceftriaxone Summary of Product Characteristics. Centre Belge d'Information Pharmacothérapeutique (C.B.I.P.asbl). Available from: http://www.cbip.be Last updated: 2015 — http://www.cbip.be
- See also: Méropénème. Meropenem Summary of Product Characteristics. Centre Belge d'Information Pharmacothérapeutique (C.B.I.P.asbl). Available from: http://www.cbip.be Last updated: 9-1-2014 — http://www.cbip.be
- See also: Temocilline. Temocillin Summary of Product Characteristics. Centre Belge d'Information Pharmacothérapeutique (C.B.I.P.asbl). Available from: http://cbip.be/ Last updated: 2014 — http://www.cbip.be